CLINICAL TRIAL: NCT02642757
Title: Effectiveness of a Brief Intervention for Reducing the Alcohol Use in Risky Users Delivered by Paramedics in Primary Care
Brief Title: Alcohol Brief Counseling in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-214; SM14I0033 (Other Grant/Funding Number: FONIS Chile)
Record Dates: First submitted 2015-12-28; First posted 2015-12-30 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Alcohol Drinking
Keywords: alcohol drinking; hazardous alcohol use; risky alcohol consumption; heavy alcohol consumption
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief intervention (Experimental): AUDIT brief intervention
  Interventions: Behavioral: AUDIT brief intervention; Other: Pamphlet on alcohol use
- Control group (Sham Comparator): Pamphlet on alcohol use
  Interventions: Other: Pamphlet on alcohol use

INTERVENTIONS:
Behavioral: AUDIT brief intervention — Intervention will be provided following the Chilean ministry of health implementation manual on the AUDIT associated brief intervention. The pamphlet on alcohol use will be provided to participants.
  Arms: Brief intervention
Other: Pamphlet on alcohol use — Only the pamphlet on alcohol use will be provided (the same received by participants on the intervention group). This is not an active intervention based on the current literature.

SUMMARY:
This study evaluates the effectiveness of a brief intervention for the reduction of alcohol use among risky alcohol users in primary care delivered by paramedics. Half of the participants will receive a brief intervention and half will receive written guidelines on safe alcohol use.

DETAILED DESCRIPTION:
Randomized controlled trial with a pragmatic emphasis undertaken in real world primary care.

The brief intervention has been designed and piloted by the mental health team at the Chilean ministry of health, as also the written support material. This intervention is the same that is being implemented national wide.

The implementation will include training of the paramedics, and then an accreditation session with a simulated participant in a double sided mirror.

Randomization will take place on site using a opaque envelope. The sequence will be keep on site in a secured box.

Data will be registered by the same person delivering the intervention and kept safe at the clinical sites. Once a month the data will be physically transferred to the operational center at the San Joaquin site of the Catholic University of Chile.

Bimonthly visits will be performed to the centers by a member of the team to assure that the protocol is being followed and data audit.

The participants will receive an economical incentive for the follow up visit. Participants will be reached throw telephone at least twice to schedule that visit. If not possible, a telephonic outcome assessment or a domiciliary visit will be performed to minimize the lost in follow up.

ELIGIBILITY:
Inclusion Criteria:

* AUDIT score between 8 and 15
* Able to read
* Haven't received a similar intervention in the last 3 months

Exclusion Criteria:

* Clients in treatment for alcohol use disorder
* Alcohol use treatment seekers
* Pregnant woman
* Severe physical or psychiatric pathology not stable

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 342 (Actual)
Dates: Start 2015-12-15; Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
AUDIT score | 6 months post brief intervention
  Total of questions 1 to 10 (minimum 0, maximum 40)

SECONDARY OUTCOMES:
AUDIT-C score | 6 months post brief intervention
  Total of questions 1 to 3 (minimum 0, maximum 12)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Barticevic, MD, Principal Investigator — Instructor Professor
Locations (5):
- Chile (5):
  - CESFAM San Alberto Hurtado, Santiago, Puente Alto
  - CESFAM Madre Teresa de Calcuta, Santiago, Puente Alto
  - CESFAM Barros Luco, Santiago, San Miguel
  - CESFAM Recreo, Santiago, San Miguel
  - CESFAM Juan Pablo II, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barticevic NA, Poblete F, Zuzulich SM, Rodriguez V, Quevedo D, Sena BF, Bradshaw L. A Health Technician-delivered Brief Intervention linked to AUDIT for reduction of alcohol use in Chilean primary care: a randomized controlled trial. Addict Sci Clin Pract. 2021 Jun 15;16(1):39. doi: 10.1186/s13722-021-00248-4. PMID 34130748